CLINICAL TRIAL: NCT06208540
Title: Persistent Olfactory and Gustatory Dysfunctions Due to Different SARS-CoV-2 Variants: Clinical Characteristics and Treatment
Brief Title: Clinical Characteristics and Treatment of Anosmia and Ageusia Due to SARS-CoV2 Variants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sherifa Ahmed Hamed (Other)
Responsible Party: Sponsor-Investigator, Sherifa Ahmed Hamed, Professor of Neurology, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-FM-covid-00325_2021
Record Dates: First submitted 2024-01-11; First posted 2024-01-17 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Post-covid-19 Persistent Smell and Taste Disorders
Keywords: COVID-19; SARS-CoV-2; variants of concern; variants of interest; Alpha strain; Delta strain; Omicron strain; Predelta period; Delta period; Omicron and its variants period
MeSH Terms: conditions — Taste Disorders; COVID-19 | interventions — cerebrolysin; Smell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients group (with interventional treatment) (Active Comparator): Patients with persistent smell and taste disorders and treated with cerebrolysin
  Interventions: Drug: Cerebrolysin; Other: olfactory and gustatory trainings
- Control (Placebo Comparator): Patients with persistent smell and taste disorders but untreated with cerebrolycin (no intervention)
  Interventions: Other: olfactory and gustatory trainings

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin Dose:5 ml ampoule (1ml contains 215.2 mg cerebrolysin) once daily through intramuscular injection five times per week, for a total of 20 treatments (for 4 weeks), after which the cycle was repeated again for at least 6 weeks till a maximum of 24 weeks.
  Other Names: Active arm
  Arms: Patients group (with interventional treatment)
Other: olfactory and gustatory trainings — olfactory and gustatory trainings using oils of strong odors for the same time frame as for the drug intervention
  Other Names: controls

SUMMARY:
The SARS-CoV-2 pandemic has consisted of multiple surges of infection because of continuous viral mutations. The WHO and CDC have defined the main SARS-CoV-2 variants based on international and national data for the circulation of SARS-CoV-2 into at least 4 waves. Studies from different parts of the world have demonstrated significant variations in the clinical manifestations of viral infection in relation to different SARS-CoV-2 variants. They also indicated that the current high levels of population immunity, due to prior infection and/or vaccination, have been associated with a vastly decreased overall risk of severe disease. Anosmia (with or without ageusia) was identified as a hallmark of COVID-19 early in the pandemic (ancestral Wuhan strain, alpha and delta variants), with a prevalence of ~60%. Prolonged olfactory disorders, lasting ≥6 months to years, has been reported in ~35-40% of infected individuals. However, studies reported that olfactory and gustatory disorders were less frequent with Omicron variants compared to pre-omicron variants. It has been indicated that SARS-CoV-2 can cause destruction, disorganization and molecular changes in the nasal olfactory neuroepithelium resulting in loss and distortion of the sense of smell. There are several trials to treat these persistent disorders but none has shown significant positive results except ours (Hamed et al., Expert Review of Clinical Pharmacology 2023;16(12):1261-1276 DOI: 10.1080/17512433.2023.2282715). Hamed et al. reported that cerebrolycin, a commercially available multimodal neurotropic factor, has the ability to cure at least 60% (100% complete and persistent recovery) of post-covid-19 persistent olfactory and gustatory dysfunctions. This drug is available in the market of at least 75 countries since 1996 and easily dispensed from local pharmacies after doctors prescriptions. It is used for treatment of many disorders of the central and peripheral nervous systems. This could be due to its ability to promote neurogenesis and remodeling of olfactory and gustatory neurons.

DETAILED DESCRIPTION:
The diminished senses of smell (or hyposmia/anosmia) and taste (or hypogeusia/ageusia) have been commonly reported after infection by ancestral Wuhan, alpha and delta strains of the SARS-CoV-2 virus in ≥ 60% of patients. Persisted dysfunctions (deficits and distortions), lasting for months to years, were also reported in ~40%.

The SARS-CoV-2 pandemic has different waves of infection because of the dynamic viral mutations. The first wave (ancestral Wuhan strain) has been defined as the period from approximately the last week of February 2020 to the first Week of February 2021; the second wave (Alpha variant) started from approximately week 7 of February 2021 to July 2021; the third wave (Delta variant) was the period from approximately August 2021 to December 2021; and the fourth wave (Omicron and its subvariants) was the period from approximately January 2022 to December 2023 and after. These Viral strains were also categorized according to the main variants and their subvariants based on the viral pathogenicity and transmissibility, the clinical manifestations, immunity and response to vaccination. Studies from different parts of the world reported less severe viral manifestations in the periods of omicron strain and its subvariants compared to the pre-omicron years of the pandemic. They also reported less frequent involvement of olfactory and gustatory systems with omicron and its subvariants compared to previous viral variants (alpha and delta).

Experimental studies strongly indicated that post-covid olfactory and gustatory disorders are due to peripheral damage of the sensory neuroepithelia (olfactory and gustatory) and their disorganization by severe viral infection and its immune mediated pathology.

In general, the characterization of the prevalence and clinical manifestations and risk variables of olfactory and gustatory complications of different SARS-CoV-2 variants is unclear. furthermore, the treatment of these prolonged complications is still aworldwide challenge. Detailed search in clinical trials' websites, for example: WHO International Clinical Trials Registry Platform (ICTRP Search Portal-WHO; https://trialsearch.who.int/), Cochrane ENT Trials Register (https://ent.cochrane.org), Ovid Embase (https://tools.ovid.com), ClinicalTrials.gov, Medfind (https:// medfind.in), Web of Science, PubMed and Scopus, demonstrated that there is only a completed and published trial which showed promising positive and maintained results (Hamed et al., 2023). In this trial, the authors concluded that cerebrolysin, a commercially available multimodal neurotropic factor, had fast, promising, and constant effect, with cure rate of >/+ 60%. This could be due to its ability to initiate and enhance neuronal regeneration, reorganization and remodeling of sensory neuroepithelia.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults with sudden hyposmia/anosmia and/or hypoageusia/ageusia during COVID-19 pandemics (2020-2024).
* Persisting symptoms were defined as disorders lasting ≥6 months.
* Cooperation during objective evaluation
* compliance to drug treatment or olfactory and gustatory trainings for at least 8 weeks.

Exclusion Criteria:

* Prior neurological, medical or psychiatric disease which are known as a cause of progressive olfactory or gustatory dysfunction
* Nasal congestion
* Nasal polyps
* Surgery or head trauma or radiation for head and neck cancers as may result in injury to the nerves that control smell
* Exposure to toxic chemicals (such as pesticides and solvents) Cocaine or other drug abuse
* Lack of compliance to drug treatment or olfactory and gustatory trainings for at least 8 weeks.
* Lack of cooperation to complete the objective testings.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
subjective evaluation | Baseline
  It included data collection of demographic, general and systemic clinical and treatment characteristics of patients infected by different SARS-CoV-2 variants. it also included the smell and taste questionnaire component of the National Health and Nutrition Examination Survey (NHNES).The dominant viral variant was defined according to the period of the development of viral manifestations including olfactory and gustatory disorders. We defined pre-delta period as February 2020 to end of May 2021; delta period as first of June 2021 till the end of December 2021; Omicron variant and its subvariants period as early in January 2022 till the end of the recruitment period.
Objective evaluation | Baseline
  It included application of modified Arabic translated and validated sniffin' odor, taste and flavor identification tests were used for objective evaluations. We used 16 different odorants which are well-known for our population. According to the results, patients were classified as normosmic (score: 12-16), hyposmic (score: 9-11) or anosmic (score: equal or less than 8). Flavor identification test was done using the same recipes as in olfactory identification test. Taste identification test was done using a five known tastants which represented the five base taste sensations (salty, sweet, bitter, sour and Umami". Answers used for the result of this test was either correct or incorrect.

SECONDARY OUTCOMES:
The Globas Rating for smell (GRS) | after 6, 8, 12, 16, 20 and 24 weeks from baseline
  It is a single-item, global rating that asks the patient to rate his current sense of smell as follow: excellent, very good, good, fair, poor or absent
The Globas Rating for taste (GRT) | after 6, 8, 12, 16, 20 and 24 weeks from baseline
  it is a single-item, global rating that asks the patient to rate his current sense of taste as follow: excellent, very good, good, fair, poor or absent
Objective re-evaluation | After 6, 8, 10, 12, 16, 20 and 24 weeks from baseline
  Sniffin' odor, taste and flavor identification tests as described in the previous section.

CONTACTS AND LOCATIONS:
Overall Officials: Sherifa A Hamed, Principal Investigator — Assiut University, Faculty of Medicine, Hospital of Neurology, Neurosurgery and Psychiatry
Locations (2):
- Egypt (2):
  - Assiut University Hospitals, Faculty of Medicine, Hospital of Neurology, Neurosurgery and Psychiatry, Assiut University Hospital, Assiut, Egypt, Asyut
  - Assiut University, Faculty of Medicine, Hospital of Neurology, Psychiatry and Neurosurgery, Asyut

IPD SHARING:
Plan to Share IPD: Yes
http://orcid.org/0000-0002-1441-3530
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 4-6 months
Access Criteria: The published work
URL: http://orcid.org/0000-0002-1441-3530

REFERENCES:
- [Result] Hamed SA, Ahmed MAA. The effectiveness of cerebrolysin, a multi-modal neurotrophic factor, for treatment of post-covid-19 persistent olfactory, gustatory and trigeminal chemosensory dysfunctions: a randomized clinical trial. Expert Rev Clin Pharmacol. 2023 Jul-Dec;16(12):1261-1276. doi: 10.1080/17512433.2023.2282715. Epub 2023 Dec 9. PMID 37950370
- [Result] Hamed SA. Post-COVID-19 persistent olfactory, gustatory, and trigeminal chemosensory disorders: definitions, mechanisms, and potential treatments. World J Otorhinolaryngol. 2023;10(2):4-22. doi: 10.5319/wjo.v10.i2.448
- [Result] Taquet M, Sillett R, Zhu L, Mendel J, Camplisson I, Dercon Q, Harrison PJ. Neurological and psychiatric risk trajectories after SARS-CoV-2 infection: an analysis of 2-year retrospective cohort studies including 1 284 437 patients. Lancet Psychiatry. 2022 Oct;9(10):815-827. doi: 10.1016/S2215-0366(22)00260-7. Epub 2022 Aug 17. PMID 35987197
- [Result] Yau JWK, Lee MYK, Lim EQY, Tan JYJ, Tan KBJC, Chua RSB. Genesis, evolution and effectiveness of Singapore's national sorting logic and home recovery policies in handling the COVID-19 Delta and Omicron waves. Lancet Reg Health West Pac. 2023 Jun;35:100719. doi: 10.1016/j.lanwpc.2023.100719. Epub 2023 Mar 2. PMID 37360873
- [Result] Micheletti C, Medori MC, Dhuli K, Maltese PE, Cecchin S, Bonetti G, Fioretti F, Assoni L, Calzoni A, Praderio A, De Angelis MG, Donato K, Arabia G, Lorusso L, Manganotti P, Capelli E, Marceddu G, Bertelli M, Nodari S. Linking pathogenic and likely pathogenic gene variants to long-COVID symptoms. Eur Rev Med Pharmacol Sci. 2023 Dec;27(6 Suppl):20-32. doi: 10.26355/eurrev_202312_34686. PMID 38112945
- [Result] Velavan TP, Ntoumi F, Kremsner PG, Lee SS, Meyer CG. Emergence and geographic dominance of Omicron subvariants XBB/XBB.1.5 and BF.7 - the public health challenges. Int J Infect Dis. 2023 Mar;128:307-309. doi: 10.1016/j.ijid.2023.01.024. Epub 2023 Jan 19. No abstract available. PMID 36681145
- [Result] Hamed SA, Kamal-Eldeen EB, Ahmed MAA. Evaluation of children and adults with post-COVID-19 persistent smell, taste and trigeminal chemosensory disorders: A hospital based study. World J Clin Pediatr. 2023 Jun 9;12(3):133-150. doi: 10.5409/wjcp.v12.i3.133. eCollection 2023 Jun 9. PMID 37342446